CLINICAL TRIAL: NCT04876651
Title: A Multinational, Multicenter, Prospective, Randomized, Controlled, Open Label Phase 3 Study With Best Standard of Care With and Without 177Lu-DOTA-rosopatamab for Patients With PSMA Expressing Metastatic Castration-resistant Prostate Cancer Progressing Despite Prior Treatment With a Novel Androgen Axis Drug
Brief Title: The Present Study Aims to Compare Patients Who Receive the Investigational Product (177Lu-DOTA-rosopatamab) Plus Standard of Care, in Comparison to Standard of Care Only
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Telix Pharmaceuticals (Innovations) Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Telix Pharmaceuticals (Innovations) Pty Limited (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 177Lu-TLX591-002
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Metastatic Prostate Cancer
Keywords: prostate cancer; 177Lu-DOTA-TLX591; progression free survival; overall survival; safety; gallium-68 labeled PSMA-11 (68Ga-PSMA-11) PET/CT Scan; novel androgen axis drug
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Approximately 387 eligible patients will be randomized to one of two groups in a 2:1 ratio to receive one of the following treatments:
  * Group A: Two single intravenous (IV) injections of 76 mCi each (equivalent to a 45 mCi/m2 dose in a standard 1.7m2 individual) of 177Lu-DOTA- rosopatamab, given 14 days apart, plus best SoC
  * Group B: Best SoC.
  Additionally, up to 10 patients, in New Zealand only, will be recruited for evaluation of biodistribution and dosimetry of 177Lu- DOTA-TLX591(m17 allotype) in combination with the SoC. These patients will receive two single intravenous (IV) injections of 76 mCi (±10%) each (equivalent to a 45 mCi/m2 dose in a standard 1.7m2 individual) of 177Lu-DOTA-TLX591 (m17), given 14 days apart, plus best SoC (abiraterone/prednisolone or enzalutamide or docetaxel). After the first dose, the patients will undergo single-photon emission computerized tomography/computerized tomography (SPECT/CT).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Two single intravenous (IV) injections of 76 mCi each (equivalent to a 45 mCi/m2 dose in a standard 1.7m2 individual) of 177Lu-DOTA- rosopatamab, given 14 days apart, plus best Standard of Care
  Interventions: Other: 177Lu-DOTA-rosopatamb
- Group B (Active Comparator): Participants will receive the Standard of Care
  Interventions: Drug: Standard of Care
- Biodistribution and Dosimetry Sub-Study (Experimental): Two single intravenous (IV) injections of 76 mCi each (equivalent to a 45 mCi/m2 dose in a standard 1.7m2 individual) of 177Lu-DOTA- rosopatamab, given 14 days apart, plus best Standard of Care
  Interventions: Other: 177Lu-DOTA-rosopatamb

INTERVENTIONS:
Other: 177Lu-DOTA-rosopatamb — Two single intravenous (IV) injections of 76 mCi each (equivalent to a 45 mCi/m2 dose in a standard 1.7m2 individual) of 177Lu-DOTA- rosopatamab, given 14 days apart, plus best SoC
  Other Names: 177Lu-TLX591
  Arms: Biodistribution and Dosimetry Sub-Study; Group A
Drug: Standard of Care — enzalutamide or abiraterone [+ prednisone/prednisolone)] or docetaxel
  Arms: Group B

SUMMARY:
This multinational, multicenter, prospective, randomized, controlled, open label Phase 3 study is designed to investigate and confirm the benefits and risks associated with the PSMA-targeted antibody, 177Lu DOTA rosopatamab administered together with Standard of Care (SoC), as compared to the best SoC alone. The phase 3 will be conducted in patients with metastatic castration-resistant PC (mCRPC) that expresses PSMA and has progressed despite prior treatment with a novel androgen axis drug (NAAD).

DETAILED DESCRIPTION:
This multinational, multicenter, prospective, randomized, controlled, open label Phase 3 study is designed to investigate and confirm the benefits and risks associated with 177Lu DOTA rosopatamab administered together with SoC, as compared to the best SoC alone, in patients with PSMA-positive, metastatic castration-resistant PC (mCRPC) that has progressed despite prior treatment with a novel androgen axis drug (NAAD).

PSMA positivity will be defined by gallium-68 labeled PSMA-11 (68Ga-PSMA-11) positron emission tomography/computerized tomography (PET/CT) as at least one site of metastatic disease with intensity significantly greater than normal liver (i.e., standardized uptake value [SUV] max at least 1.5 times SUV of normal liver.

Approximately 392 eligible adult male will be part of this study. 387 patients will be randomized to one of two groups in a 2:1 ratio to receive one of the treatments below. 5 participants in New Zealand will be enrolled into a sub-study.

* Group A: Two single intravenous (IV) injections of 76 mCi each (equivalent to a 45 mCi/m2 dose in a standard 1.7m2 individual) of 177Lu-DOTA- rosopatamab, given 14 days apart, plus best SoC
* Group B: Best SoC.

In parallel to this, 5 participants in New Zealand site, will be enrolled into a sub-study to investigate the biodistribution, pharmacokinetics and dosimetry of 177Lu-DOTA-TLX591(m17). Participants will receive two doses of 177Lu-DOTA-TLX591(m17), 14 days apart.

Screening procedures will take up to 28 days prior to enrollment and randomization. Only patients with PSMA-positive metastatic PC and meeting all other inclusion/exclusion criteria were randomized in a 2:1 ratio to Group A or B OR allocated to Sub-study in New Zealand.

Participants in Group A or B will participate in the study for up to 5 years. During this period the participants will undergo imaging procedures approximately every 6-8 weeks until progression.

Participants in the sub-study will participate in the study up to 23 days. During this period participants will receive two doses of 177Lu-DOTA-TLX591(m17), 14 days apart, and undergo SPECT/CT imaging and blood collection for Pharmacokinetics at days 1,2,5,8, 13 and 15.

For all patients, the best SoC will be determined by the Principal Investigator (PI) and the medication will be provided until progression.

ELIGIBILITY:
Inclusion Criteria:

1. Be a male, at least 18 years old, with metastatic adenocarcinoma of the prostate defined by histological / pathological confirmation of PC.
2. Be of ECOG Performance Status 0, 1, or 2 and have an estimated life expectancy of ≥6 months.
3. Have metastatic disease (≥1 metastatic lesions present on baseline CT, MRI, or bone scan imaging).
4. Have castration-resistant PC (defined as disease progressing despite castration by orchiectomy or ongoing use of luteinizing hormone-releasing hormone [LHRH]) and must have a castrate level of serum/plasma testosterone (<50 ng/dL or <1.7 nmol/L).
5. In the mCRPC setting, must have received a minimum of 12 weeks of prior therapy with a NAAD, either enzalutamide or abiraterone plus prednisone.
6. Should have received one line of prior taxane therapy or have refused or be ineligible for taxanes
7. Have a disease that is progressing at study entry, despite a castrate testosterone level (<50 ng/dL or <1.7 nmol/L), by the demonstration of at least one of the following:

   1. Rising PSA values done in sequence at least 1 week apart and with a minimal starting value of 2.0 ng/mL.
   2. Progressive disease or new lesion(s) in the viscera or lymph nodes as per RECIST1.1 or in bone as per Prostate Cancer Working Group 3 [PCWG3; Scher et al., 2016]). Any ambiguous results are to be confirmed by other imaging modality (e.g., CT or MRI scan).
8. Have disease that is PSMA positive, as demonstrated by a 68Ga-PSMA11 PET/CT scan and confirmed as eligible by the Sponsor's central reader (patient must have at least one site of metastatic disease with SUVmax ≥1.5 times the SUV of normal liver). If the disease meets the criteria for PSMA positivity, but there is one or more soft tissue lesion of ≥ 2 cm that is not PSMA positive, then the patient is to be excluded on the grounds that there is substantial disease which might not respond to the therapy.
9. Must have recovered to ≤ Grade 2 from all clinically significant toxicities related to prior therapies (i.e., surgery, local radiotherapy, NAAD, chemotherapy, etc.).
10. Can be receiving a bisphosphonate or denosumab regimen provided that the patient has been receiving and tolerating this treatment for ≥30 days prior to randomization.
11. Have adequate organ function at Screening:

    a. Bone marrow: i. Platelets ≥150×109/L. ii. Absolute neutrophil count >1.5×109/L. iii. Hemoglobin ≥10g/dL (no red blood cell transfusion in the previous 4 weeks).

    b. Liver function: i. Total bilirubin < 1.5×the upper limit of normal (ULN). For patients with known Gilbert's Syndrome <3×ULN is permitted. ii. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) <3×ULN OR <5×ULN for patients with liver metastases. c. Renal function: i. Serum/plasma creatinine <1.5×ULN or creatinine clearance ≥50 mL/min determined using the Cockcroft & Gault formula.
12. Have the capacity to understand the study and be able and willing to comply with all protocol requirements.
13. Patients must comply with the radiation protection rules (including hospital admissions and isolation) that are used by the treating institution in order to protect their contacts and the general public, especially if a female partner of the patient is or could be pregnant.
14. Must agree to practice adequate precautions to prevent pregnancy in a partner and to avoid potential problems associated with radiation exposure to the unborn child (Refer to Clinical Trials Facilitation Group, 2020: Recommendations related to contraception and pregnancy testing in clinical trials Version 1.1, CTFG, 2020).

Exclusion Criteria:

1. Are unable to understand or are unwilling to sign a written informed consent document or to follow investigational procedures in the opinion of the Investigator.
2. Have PC associated with pathological findings consistent with small cell or any histology other than adenocarcinoma of the prostate. If there are minor elements of neuroendocrine histology, this is acceptable.
3. Uncontrolled pain.
4. Diagnosed with other malignancies that are expected to alter life expectancy or may interfere with disease assessment. However, patients with a prior history of malignancy that has been adequately treated and who have been disease-free for more than 3 years are eligible, as are patients with adequately treated non-melanoma skin cancer, and superficial bladder cancer.
5. Are at increased risk of hemorrhage or bleeding, or with a recent history of a thrombolytic event (e.g., deep vein thrombosis [DVT]/ pulmonary embolism [PE]) and have been administered long-term anti-coagulant or anti-platelet agents.
6. Have received prior treatment with monoclonal antibody (mAb) J591 or HuJ591 or any other PSMA targeted therapy.
7. Have known allergies, hypersensitivity, or intolerance to the investigational drug or its excipients.
8. Have received prior systemic anti-cancer therapy (e.g., chemotherapy, immunotherapy, or biological therapy) and/or radiation therapy within 4 weeks of randomization OR if any significant AEs have not resolved to National Cancer Institute (NCI) AE Criteria ≤2; OR are receiving other concurrent cytotoxic chemotherapy, immunotherapy, radioligand therapy, or investigational therapy.
9. Have received prior treatment with radioisotopes, including but not limited to: 89Strontium, 153Samarium, 186Rhenium, 188Rhenium, 223Radium, or hemi-body irradiation within 6 months prior to randomization.
10. Have received other investigational therapy within 4 weeks of randomization.
11. Have known brain metastases or hepatic metastases.
12. Have a history of seizure and/or stroke within past 6 months.
13. Have clinical or radiologic findings indicative of impending cord compression or experience symptomatic cord compression.
14. Have a serious active or sub-clinical infection or angina pectoris (New York Heart Association [NYHA] Class III or IV), significantly prolonged QT interval or other serious illness(es) involving the cardiac, respiratory, central nervous system, renal, hepatic or hematological organ systems, which might impair the ability to complete this study or could interfere with determination of causality of any adverse effects experienced in this study, or which require treatment that could interact with study treatment, particularly with enzalutamide.
15. Have received treatment with any PARP inhibitors (i.e., Olaparib) or with any platinum based anti-neoplastic drugs.
16. Have a known alteration in breast cancer genes (BRCA) BRCA1, BRCA2, or Ataxia Telangiectasia Mutated Gene (ATM) gene and are eligible to receive Olaparib therapy according to their institution's SoC

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Estimated)
Dates: Start 2023-08-29 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of radiographic progression-free survival (rPFS) | Day 1 to 5 years after two administrations of 177Lu-DOTA-rosopatamab
  Radiographic progression-free survival (rPFS) defined as the time from randomization to disease progression confirmed by central independent radiology review according to RECIST 1.1 (for soft tissue disease) and/or PCWG3 criteria (for bone disease), or death (whichever occurs first).

SECONDARY OUTCOMES:
Overall survival | Day 1 to 5 years after two administrations of 177Lu-DOTA-rosopatamab
  Overall survival (OS), determined from randomization, until death from any cause
Tumour objective response rate (ORR) | Day 1 to 5 years after two administrations of 177Lu-DOTA-rosopatamab
  Tumor response in terms of objective response rate (ORR) (malignant soft tissue response and overall radiological response [malignant soft tissue response by RECIST 1.1 and overall radiological response by RECIST 1.1 and PCWG3]).
Time to a first Symptomatic Skeletal Event (SSE) | Day 1 to 5 years after two administrations of 177Lu-DOTA-rosopatamab
  Time to a first SSE, defined as the use of external beam radiation to relieve bone pain, or occurrence of a new symptomatic pathological fracture (vertebral or non-vertebral), or occurrence of spinal cord compression, or tumor-related orthopedic surgical intervention
Progression-free survival | Day 1 to 5 years after two administrations of 177Lu-DOTA-rosopatamab
  PFS defined as the time from randomization to disease progression confirmed by radiology, clinical or PSA progression, or death (whichever occurs first).
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Day 1 to 5 years after two administrations of 177Lu-DOTA-rosopatamab
  Assessment of AEs graded by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0, vital signs (systolic and diastolic blood pressures, respiratory rate, pulse rate, and body temperature), ECGs, and evaluation of laboratory parameters (biochemistry, hematology, coagulation, and urinalysis).
Adverse events of special interest (AESI) | Day 1 to 5 years after two administrations of 177Lu-DOTA-rosopatamab
  Assessment of any Grade 4 hematological abnormalities and bleeding events and Symptomatic skeletal events (SSE), defined as the use of external beam radiation to relieve bone pain, or occurrence of a new symptomatic pathological fracture (vertebral or non-vertebral), or occurrence of spinal cord compression, or tumor-related orthopedic surgical intervention.
Health-related quality of life by ECOG | Day 1 to 5 years after two administrations of 177Lu-DOTA-rosopatamab
  Quality of Life is to be evaluated using the Eastern Cooperative Oncology Group (ECOG) Performance Scale- From 0 (fully active) to 5 (dead).
Health-related quality of life by FACT-P | Day 1 to 5 years after two administrations of 177Lu-DOTA-rosopatamab
  The Functional Assessment of Cancer Therapy-Prostate (FACT-P) evaluates the physical well-being, social/family well-being, emotional well-being and functional well-being), the results range from "not at all" to "Very much"
Health-related quality of life by BPI-SF | Day 1 to 5 years after two administrations of 177Lu-DOTA-rosopatamab
  The Brief Pain Inventory - Short Form (BPI-SF) where the results vary from 1-4 (mild pain), 5-6 (Moderate pain) and 7-10 (severe pain)
Health-related quality of life by EQ-5D-5L | Day 1 to 5 years after two administrations of 177Lu-DOTA-rosopatamab
  The EQ-5D-5L where the results vary from 1 (no problems) to 5 (extreme problems/unable to do)
Health-related quality of life by EORTC/QQ-C30 | Day 1 to 5 years after two administrations of 177Lu-DOTA-rosopatamab
  The European Organisation for Research and Treatment of Cancer (EORTC) Core Quality of Life Questionnaire (QLQ-C30) questionnaire - result is calculated from the mean of 13 of the 15 QLQ-C30 scales (Physical Functioning+ Role Functioning+ Social Functioning+ Emotional Functioning+ Cognitive Functioning+ Fatigue+ Pain+ Nausea_Vomiting+ Dyspnoea+ Sleeping Disturbances+ Appetite Loss+ Constipation+ Diarrhoea) ranging from "not at all" to "Very much"
Assessment of changes in prostate specific antigen (PSA) | Day 1 to 5 years after two administrations of 177Lu-DOTA-rosopatamab
  Percentage change from baseline in PSA level, PSA response, and PSA response duration
Time to radiographic soft tissue progression (TTSTP) | Day 1 to 5 years after two administrations of 177Lu-DOTA-rosopatamab
  Time to radiographic soft tissue progression (TTSTP) defined as time from randomization to radiographic soft tissue progression according to RECIST 1.1 (for soft tissue disease).
Biochemical response as indicated by PSA levels, lactate dehydrogenase (LDH) and alkaline phosphatase (ALP) levels | Day 1 to 5 years after two administrations of 177Lu-DOTA-rosopatamab
  Percentage change from baseline in PSA level, PSA response, and PSA response duration and percentage change from baseline in blood LDH/ALP levels.
Development of anti-drug antibodies (ADA) to 177Lu-DOTA-TLX591 | Day 1 to 5 years after two administrations of 177Lu-DOTA-rosopatamab
  A blood test to check if antibodies are formed against the study drug, and how much of the antibodies is formed and if it is enough to neutralize the study drug. ADA can reduce or neutralise the drug's effectiveness as the body tries to neutralize the drug.
Titer of anti-drug antibodies (ADA) to 177Lu-DOTA-TLX591 | Day 1 to 5 years after two administrations of 177Lu-DOTA-rosopatamab
  The concentration (ug/mL) of anti-drug antibodies (ADA) to 177Lu-DOTA-TLX591
Duration of positiveness in the development of anti-drug antibodies (ADA) to 177Lu-DOTA-TLX591 | Day 1 to 5 years after two administrations of 177Lu-DOTA-rosopatamab
  In case of DA positiveness, this will analise how long the ADA positiveness is measured in the study samples.
Neutralizing anti-drug antibodies (NAb) to 177Lu-DOTA-TLX591 | Day 1 to 5 years after two administrations of 177Lu-DOTA-rosopatamab
  How many study samples have been positive (rate) for neutralizing anti-drug antibodies (NAb) to 177Lu-DOTA-TLX591. NAb can neutralize the biological drugs and decrease the drug's efficacy and increase its clearance, resulting in patient secondary unresponsiveness.
To determine whole body biodistribution (BD) of administered activity 177Lu-DOTATLX591(m17) | Day 1 to day 23 after two administrations of 177Lu-DOTA-rosopatamab
  Evaluate whole body and organs imagining positivity for administered 177Lu-DOTATLX591 (m17)
To determine organ radiation dosimetry of tracer levels of administered activity 177Lu-DOTATLX591(m17) | Day 1 to day 23 after two administrations of 177Lu-DOTA-rosopatamab
  Evaluate organs absorbed radiation doses of administered 177Lu-DOTATLX591 in PSMA expressing tumours as determined by suitable tumour-to-heathy tissue ratios and residence times.
To determine pharmacokinetics (PK) of administered activity 177Lu-DOTATLX591 | Day 1 to day 23 after two administrations of 177Lu-DOTA-rosopatamab
  Measure whole blood radioactive concentration at each timepoint to determine the radiation PK curve.
Demonstrate comparability of whole body biodistribution dosimetry of the 177Lu-DOTA-TLX591 | Day 1 to day 23 after two administrations of 177Lu-DOTA-rosopatamab
  Qualitative comparison measured in SUV (Standardized Uptake Value) of whole-body biodistribution between 177Lu-DOTA-TLX591 from ProstACT-SELECT participants (NCT04786847) and this study's participants
Demonstrate comparability of organ uptake dosimetry of the 177Lu-DOTA-TLX591 | Day 1 to day 23 after two administrations of 177Lu-DOTA-rosopatamab
  Qualitative comparison measured in SUV (Standardized Uptake Value) of organ uptake between 177Lu-DOTA-TLX591 from ProstACT-SELECT participants (NCT04786847) and this study's participants
Demonstrate organ radiation dosimetry comparability of the 177Lu-DOTA-TLX591 | Day 1 to day 23 after two administrations of 177Lu-DOTA-rosopatamab
  Qualitative comparison of organ dosimetry from ProstACT-SELECT participants (NCT04786847) and 177Lu-DOTA-TLX591 (m17 allotype)

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (5):
  - Westmead Hospital, Westmead, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Monash Health, Clayton, Victoria
  - Austin Health, Melbourne, Victoria
  - 'GenesisCare Murdoch', Murdoch, Western Australia
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No